CLINICAL TRIAL: NCT00314977
Title: Sequential vs Upfront Intensified Neoadjuvant Chemotherapy in Patients With Large Resectable and/or Locally Advanced Breast Cancer. The INTENS Study
Brief Title: Sequential vs Upfront Intensified Neoadjuvant Chemotherapy in Patients With Large Resectable or Locally Advanced Breast Cancer.
Acronym: INTENS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Collaborators: Sanofi (Industry); Amgen (Industry)
Responsible Party: Prof dr V.C.G. Tjan-Heijnen, Maastricht University Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IKO 2005-01 / BOOG 2007-02
Record Dates: First submitted 2006-04-14; First posted 2006-04-17 (Estimated); Last update posted 2010-03-18 (Estimated); Status verified 2010-03

CONDITIONS: Breast Cancer
Keywords: Large resectable breast cancer; Locally advanced breast cancer; Neoadjuvant therapy
MeSH Terms: conditions — Breast Neoplasms | interventions — Doxorubicin; Cyclophosphamide; Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental): Cycles 1-4 q 3 weeks: doxorubicin plus cyclophosphamide Cycles 5-8 q 3 weeks: docetaxel
  Interventions: Drug: Doxorubicin; Drug: Cyclophosphamide; Drug: Docetaxel
- B (Experimental): Cycles 1-6 q 3 weeks: doxorubicin, cyclophosphamide and docetaxel
  Interventions: Drug: Doxorubicin; Drug: Cyclophosphamide; Drug: Docetaxel

INTERVENTIONS:
Drug: Doxorubicin — doxorubicin (arm A:60 mg/m2) and arm B: 50 mg/m2)
  Other Names: hydroxyldaunorubicin; adriamycin
Drug: Cyclophosphamide — Cyclophosphamide: (arm A; 6000 mg/m2) an (arm B: 500 mg/m2)
  Other Names: Cytoxan; Neosar; Revimmune
Drug: Docetaxel — Docetaxel: (arm A: 100 mg/m2) and (arm B: 75 mg/m2)
  Other Names: Taxotere

SUMMARY:
2 different treatment schedules may be used for neoadjuvant chemotherapy in breast cancer using adriamycin, cyclophosphamide and taxotere. The most optimal sequence- concurrent or sequential- is however unclear. The aim of the study is to compare the efficacy and tolerability of neoadjuvant chemotherapy with AC followed by T(adriamycin, cyclophosphamide, taxotere) versus TAC ( with upfront T) in patient with large resectable or locally advanced breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* Women presenting with large resectable or locally advanced breast cancer (T2 ≥3 cm, T3, or T4, and/or LN positive)
* Measurable disease (breast and/or lymph nodes)
* No prior surgery other than biopsy and no prior chemotherapy or radiation therapy
* Age ≥18 years and age ≤70 years
* Karnofsky Performance score ≥70%
* Estrogen and/or progesterone receptor analysis performed on the primary tumour in the biopsy material
* In case the tumor is ER/PgR ³ 50% positive, (neo)adjuvant hormonal therapy in stead of chemotherapy should be considered (e.g. in TEAM II study)
* Her2/neu receptor analysis performed on the primary tumour in the biopsy material
* Adequate bone marrow function (within 14 days prior to registration): WBC ≥3.0 x 109/l, neutrophils ≥1.5 x 109/l, platelets ≥100 x 109/l
* Adequate liver function (within 4 weeks prior to start treatment): bilirubin ≤1.5 x upper limit of normal (UNL) range, ALAT and/or ASAT ≤2.5 x UNL, Alkaline Phosphatase ≤5 x UNL
* Adequate renal function (within 4 weeks prior to start treatment): the calculated creatinine clearance should be ≥50 mL/min
* Patients must be accessible for treatment and follow-up
* Written informed consent according to the local Ethics Committee requirements

Exclusion Criteria:

* Patients with advanced pulmonary disease of any cause (oxygen dependent)- Peripheral neuropathy > grade 2 whatever the cause
* Serious other diseases as recent myocardial infarction, clinical signs of cardiac failure or clinically significant arrythmias
* Evidence of distant metastases (M1)
* Patients with a history of breast cancer
* Patients with a history of another malignancy (except basal cell skin carcinoma and carcinoma-in-situ of the uterine cervix) within 5 years of study entry- Pregnant or lactating women, or potentially fertile women not using adequate contraception

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2006-02; Primary Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
The pathologic complete response rate to neoadjuvant chemotherapy.

SECONDARY OUTCOMES:
The delivered chemotherapy dose and dose-intensity of both chemotherapy regimens
The tolerability (grade 3/4 CTC toxicities) of both chemotherapy regimens.
The clinical responses of neoadjuvant chemotherapy correlated to pathological responses after neoadjuvant chemotherapy.
The value of breast MRI in evaluating response to neoadjuvant chemotherapy as compared to clinical palpation, ultrasound techniques and histo-pathological outcome.
The false-negative rate of the sentinel node biopsy after neoadjuvant chemotherapy.
The disease-free and overall survival after 3 and 5 years follow-up.
The relation between pCR and DFS/OS.
The feasibility of the criteria for reporting pathological tumour response in surgical breast and axillary node resection specimens.
The prognostic and predictive value of tumour- and molecular markers, including ER, PgR, c-erbB2, microarray and other tumour characteristic analyses.

CONTACTS AND LOCATIONS:
Overall Officials: V.C.G. Tjan-Heijnen, Principal Investigator — AZM Maastricht
Locations (24):
- Netherlands (24):
  - Jeroen Bosch Ziekenhuis, 's-Hertogenbosch
  - Onze Lieve Vrouwe Gasthuis, Amsterdam
  - Rijnstate Ziekenhuis, Arnhem
  - Deventer Ziekenhuis, Deventer
  - Slingeland Hospital, Doetinchem
  - Catharina Ziekenhuis, Eindhoven
  - St. Anna Hospital, Geldrop
  - St. Jansdal Ziekenhuis, Harderwijk
  - Atrium Medisch Centrum, Heerlen
  - Elkerliek Ziekenhuis, Helmond
  - Spaarne Ziekenhuis, Hoofddorp
  - Leids Universitair Medisch Centrum (LUMC), Leiden
  - Academical Hospital Maastricht (AZM), Maastricht
  - St. Antonius Hospital, Nieuwegein
  - Canisius Wilhelmina Ziekenhuis, Nijmegen
  - Radboud University Medical Centre, Nijmegen
  - Waterland Hospital, Purmerend
  - Maasland Hospital, Sittard
  - HAGA Ziekenhuis, The Hague
  - St. Elisabeth Ziekenhuis, Tilburg
  - Mesos Medisch Centrum, Utrecht
  - UMC Utrecht, Utrecht
  - Maxima Medisch Centrum, Veldhoven
  - Zaans Medical Centre, Zaandam

REFERENCES:
- [Derived] Vriens BEPJ, Vriens IJH, Aarts MJB, van Gastel SM, van den Berkmortel FWPJ, Smilde TJ, van Warmerdam LJC, van Spronsen DJ, Peer PGM, de Boer M, Tjan-Heijnen VCG; Breast Cancer Trialists' Group of the Netherlands (BOOG). Improved survival for sequentially as opposed to concurrently delivered neoadjuvant chemotherapy in non-metastatic breast cancer. Breast Cancer Res Treat. 2017 Oct;165(3):593-600. doi: 10.1007/s10549-017-4364-8. Epub 2017 Jul 3. PMID 28674765
- [Derived] Vriens BE, de Vries B, Lobbes MB, van Gastel SM, van den Berkmortel FW, Smilde TJ, van Warmerdam LJ, de Boer M, van Spronsen DJ, Smidt ML, Peer PG, Aarts MJ, Tjan-Heijnen VC; INTENS Study Group. Ultrasound is at least as good as magnetic resonance imaging in predicting tumour size post-neoadjuvant chemotherapy in breast cancer. Eur J Cancer. 2016 Jan;52:67-76. doi: 10.1016/j.ejca.2015.10.010. Epub 2015 Nov 30. PMID 26650831